CLINICAL TRIAL: NCT00941148
Title: Impact of Insulin (I.)Glargine Compared to NPH I. and to I. Detemir in Combination With Metformin on Prandial ß-cell Function and Overall Metabolic Control in Type 2 Diabetic Patients With Insufficient Metabolic Control During OAD Treatment
Brief Title: Beta-Cell Function of Insulin Glargine Compared to Neutral Protamine Hagedorn (NPH) Insuline and to Insulin Detemir in Combination With Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Prof. Thomas Forst, MD, ikfe GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANT_001; EudraCT Number: 2007-006109-26
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetic Patients; Insufficient Metabolic Control; OAD Treatment
MeSH Terms: interventions — Insulin, Isophane; Insulin Detemir; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Insulin glargine (Active Comparator): Insulin glargine, dose individually adapted to reach treatment goal (FBG < 100 mg/dL)
  Interventions: Drug: Insulin Glargin; Drug: metformin
- NPH Insulin (Active Comparator): NPH Insulin, dose individually adapted to reach treatment goal (FBG < 100 mg/dL)
  Interventions: Drug: NPH insulin; Drug: metformin
- Insulin detemir (Active Comparator): Insulin detemir, dose individually adapted to reach treatment goal (FBG < 100 mg/dL)
  Interventions: Drug: Insulin detemir; Drug: metformin

INTERVENTIONS:
Drug: Insulin Glargin
  Arms: Insulin glargine
Drug: NPH insulin
  Arms: NPH Insulin
Drug: Insulin detemir
  Arms: Insulin detemir
Drug: metformin — metformin (2000 mg/day)

SUMMARY:
The aim of the study is to show that treatment with Glargine will lead to an improvement in beta cell function especially within times of maximal beta cell stress occurring after a meal. For this reason three different standardized test meals (breakfast, lunch, dinner) will be performed and the postprandial secretion of intact proinsulin levels will be measured. These measurements will be performed with patients treated in combination with metformin and insulin glargine versus metformin plus NPH insulin (within the core study) and if significant difference is observed, with a third treatment arm with metformin plus insulin detemir.

Hypothesis is that the area under the curve (AUC) intact proinsulin levels within 2 hours after test meal dinner of metformin plus insulin glargin differs from AUC intact proinsulin levels of metformin plus NPH insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus according to the ADA criteria
* HbA1c between 6.5% and 8.5%
* Individually optimized combination therapy with metformin in combination with sulfonylurea in a stable dosage within the last 3 months
* Age between 40 and 75 years
* Fasting intact proinsulin level > 7 pmol/Land < 20 pmol/Lat screening

Exclusion Criteria:

* Type 1 Diabetes mellitus
* Pre-Treatment with insulin within the last 3 months prior to screening
* Pre-Treatment with PPARy-agonists (glitazones) within the last 3 months prior to screening
* Major micro- or macrovascular complications as judged by the investigator
* BMI > 40 kg/m²
* Hypokalemia (K < 3.5 mmol /L)
* History of drug or alcohol abuse
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures
* History of severe or multiple allergies
* Treatment with any other investigational drug within 3 months prior to screening
* Progressive fatal disease
* History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (creatinine > 1.3 mg/dL in women and > 1.7 mg/dL in men), neurological, psychiatric and/or haematological disease as judged by the investigator
* Pregnancy or breast feeding
* Sexually active women of childbearing potential not actively and consistently practicing birth control by using a medically accepted device or therapy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
postprandial dynamics of intact proinsulin secretion after standardized test meals (AUC for two hours after dinner) | 12 +/- 2 weeks

SECONDARY OUTCOMES:
AUC for intact proinsulin levels for two hours after a standardized test meal (breakfast and lunch) | 12 +/- 2 weeks
increase of intact proinsulin after breakfast (BF), lunch (LU) and dinner (DI) | 12 +/- 2 weeks
Ratio of exogenous insulin vs. endogenous insulin (measurements of glargine, NPH Insulin, detemir and human insulin levels) | 12 +/- 2 weeks
Postprandial endothelial function measured as postischaemic response in LDF measurements (after BF, LU, DI) | 12 +/- 2 weeks
Postprandial change in and AUC for hs CRP (after BF, LU, DI) | 12 +/- 2 weeks
Postprandial change in and AUC for ADMA (after BF, LU, DI) | 12 +/- 2 weeks
Postprandial increase in and AUC for glucose levels (after BF, LU, DI) | 12 +/- 2 weeks
Changes in FBG | 12 +/- 2 weeks
Changes in 8-point BG profiles | 12 +/- 2 weeks
Percentage of patients reaching the treatment goal | 12 +/- 2 weeks
Insulin dosage per kg body weight to reach treatment goal | 12 +/- 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ikfe GmbH, Clinic Department, Mainz, RLP, Germany

REFERENCES:
- [Derived] Forst T, Larbig M, Hohberg C, Forst S, Diessel S, Borchert M, Roth W, Pfutzner A. Adding insulin glargine vs. NPH insulin to metformin results in a more efficient postprandial beta-cell protection in individuals with type 2 diabetes. Diabetes Obes Metab. 2010 May;12(5):437-41. doi: 10.1111/j.1463-1326.2010.01209.x. PMID 20415692